CLINICAL TRIAL: NCT04832035
Title: Integration of Refugees With Mental Disorders Into the Public Psychotherapeutic Health Care Services - a Model Project With Trained Peers
Brief Title: Integration of Refugees Into Public Mental Health Care
Acronym: INT_REF_MH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Konstanz (Other)
Collaborators: Vivo international e.V. (Industry)
Responsible Party: Principal Investigator, Michael Odenwald, CEO psychotherapeutic outpatient clinic, leading psychologist research ward, University of Konstanz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Refugee Integration 2021
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Psychiatric Disorders From Chapters 3 and 4 of ICD10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard psychotherapeutic care + coordinated and peer supported mental health care" (Experimental): Participants receive standard psychotherapeutic care in the public healthcare system. For participants and therapists in this group standard care and additional organisational support is available which is labeled "coordinated and peer supported mental health care". This includes several additional organisational assistance components that are currently not part of the services of the public mental health care system, i.e. a coordination center, trained peers to support treatment utilisation, a support and training center for therapists, and an interpreter pool.This is Treatment as Usual plus coordination and peer support.
  Interventions: Other: "coordinated and peer supported mental health care"; Behavioral: "standard psychotherapeutic care in the public healthcare system"
- Standard psychotherapeutic care" (Other): Participants receive standard psychotherapeutic care in the public healthcare system. For participants in this group no additional organisational support is available. This is Treatment as Usual.
  Interventions: Behavioral: "standard psychotherapeutic care in the public healthcare system"

INTERVENTIONS:
Other: "coordinated and peer supported mental health care" — Health services, coordination of services, method to support utilization
  Arms: Standard psychotherapeutic care + coordinated and peer supported mental health care"
Behavioral: "standard psychotherapeutic care in the public healthcare system" — Psychotherapeutic services that are financed by the public health insurance system.

SUMMARY:
There are specific barriers to utilise psychotherapeutic services for refugees with mental health problems in the German public health care system. This study aims to evaluate additional organisational components that are hypothesised to improve service utilisation.

In a randomised controlled trial, refugees with mental health problems are identified by peers, subsequently assessed by professional staff and referred to public psychotherapeutic health services who offer standard care. Participants are assigned to care as usual or to "coordinated and peer supported mental health care"; the latter includes several additional organisational assistance components, i.e. a coordination center, trained peers to support treatment utilisation, a support and training center for therapists, and a interpreter pool. Measures include service utilisation and symptom change after 6 months. Furthermore the study evaluates whether trained peers can correctly identify participants with mental health problems.

ELIGIBILITY:
Inclusion Criteria:

* Psychiatric diagnosis from Chapters 3 and 4 of ICD10
* Participant applied for asylum in Germany
* Entry to Germany after 2012
* Participants is motivated to utilise psychotherapeutic services
* Patient speaks one of the languages in which services are offered (i.e. German, English, French, Arabic, Kurdish, Dari, Farsi, Urdu, Pashto, Tirginya, Somali)

Exclusion Criteria:

* Mental disorder that requires inpatient treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Service utilisation | 6 months after study inclusion
  Percentage of participants who utilise psychotherapeutic services
Psychiatric symptom change | assessments 6 and 12 months after study inclusion
  Self-report of psychiatric symptoms by means of questionnaires

SECONDARY OUTCOMES:
Percentage correctly identified refugees with mental health problems | two weeks
  Comparison of peer screening and expert diagnostic assessment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Konstanz, Psychotherapy Outpatient Clinic, Konstanz, Germany

IPD SHARING:
Plan to Share IPD: Undecided